CLINICAL TRIAL: NCT01325415
Title: A Single Center, Randomized, Double-blinded, Placebo-controlled, Open-label, Positive-controlled, Four-way Crossover Study to Assess the Effect of a Single Oral Dose NKTR-118 Administration on QTc Interval Compared to Placebo, Using AVELOX (Moxifloxacin) as a Positive Control, in Healthy Male Subjects
Brief Title: A Placebo-controlled Four Way Crossover Study to Asses the Effect of a Single Oral Dose of NKTR-118 on QTc Interval in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D3820C00014
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Amount of NKTR-118 in Blood; Variation in the Heart's Electrical Cycle
Keywords: Phase 1; healthy male volunteers; cross-over study; NKTR-118
MeSH Terms: interventions — naloxegol; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): NKTR-118 25 mg (1x25 mg tablet + 5x placebo tablets)
  Interventions: Drug: NKTR-118; Drug: Placebo
- B (Experimental): NKTR-118 150 mg (6x25 mg tablet)
  Interventions: Drug: NKTR-118; Drug: Placebo
- C (Placebo Comparator): NKTR-118 placebo (6x placebo tablets)
  Interventions: Drug: Placebo
- D (Active Comparator): Moxifloxacin (1 x 400 mg tablet)
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: NKTR-118 — 25 mg tablet
  Arms: A; B
Drug: moxifloxacin — 400 mg tablet
  Arms: D
Drug: Placebo — tablet
  Arms: A; B; C

SUMMARY:
The purpose of this study is to evaluate the effects on QTc interval in healthy males when administered a single dose of NKTR-118 compared with placebo and moxifloxacin. (QTc is a specific time interval that can be measured in a heart beat by taking Electrocardiogram (ECG))

DETAILED DESCRIPTION:
A Single Center, Randomized, Double-blinded, Placebo-controlled, Open-label, Positive-controlled, Four-way Crossover Study to Assess the Effect of a Single Oral Dose NKTR-118 Administration on QTc Interval Compared to Placebo, Using AVELOX (moxifloxacin) as a Positive Control, in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and weight at least 50 kg but no more than 100 kg.

Exclusion Criteria:

* Clinically significant medical history including severe allergies or a history of mental disorders or any cardiac history, history or presence of gastrointestinal, hepatic, or renal disease.
* Abnormal heart rhythm including any abnormal arrhythmias, marked sinus arrhythmias, or junctional rhythms.
* Known or suspected history of drug abuse, current smokers or those who have smoked and/or used nicotine products within 3 months prior to enrollment.
* Excessive intake of caffeine-containing products

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a single dose of NKTR-118 25 mg and 150 mg on the change in time-matched QTcF intervals compared with placebo | 30 days pre-dose through 4 treatment periods and follow up 71 days post dose.
The effect of a single dose of NKTR-118 25 mg and 150 mg on the change in time-matched QTcF intervals compared with placebo | Follow up 71 days post dose.

SECONDARY OUTCOMES:
To evaluate the effect of a single oral dose of moxifloxacin 400 mg on the changes in time-match QTcF intervals compared with placebo, which will be used as supporting data. | 30 days pre-dose through 4 treatment periods
Collect adverse events to assess the safety after dosing of NKTR-118 25mg and 150 mg in healthy male subjects. | 30 days pre-dose through 4 treatment periods
To evaluate the effect of a single oral dose of moxifloxacin 400 mg on the changes in time-match QTcF intervals compared with placebo, which will be used as supporting data. | Follow up 71 days post dose
Collect adverse events to assess the safety after dosing of NKTR-118 25mg and 150mg in healthy male subjects. | Follow up 71 days post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca, Wilmington US; David Matthews, MD, Principal Investigator — Quintiles, Overland Park Kansas US; Emilie Ramos, MD, Study Chair — AstraZeneca, Alderley Park, UK
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Gottfridsson C, Carlson G, Lappalainen J, Sostek M. Evaluation of the effect of Naloxegol on cardiac repolarization: a randomized, placebo- and positive-controlled crossover thorough QT/QTc study in healthy volunteers. Clin Ther. 2013 Dec;35(12):1876-83. doi: 10.1016/j.clinthera.2013.09.019. Epub 2013 Nov 13. PMID 24238792
- See also: D3820C00014 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1395&filename=D3820C00014_Clinical_Study_Report_Synopsis.pdf